CLINICAL TRIAL: NCT03090087
Title: The Effect of A2A Adrenoceptor Stimulation on the Diameter of Retinal Arterioles During Hypoxia in Vivo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Adenosine RVA
Record Dates: First submitted 2017-03-10; First posted 2017-03-24 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Retinal Artery Occlusion
Keywords: Diameter of retinal arteries; Adenosine; Hypoxia
MeSH Terms: conditions — Retinal Artery Occlusion; Hypoxia | interventions — regadenoson

STUDY DESIGN:
Intervention Model Description: The project will be conducted as an open controlled interventional study performed on two days separated by at least one day.
  The test persons will be randomly allocated to two groups, one group in which protocol 1 is followed by protocol 2, and the other group with the two protocols performed in the reverse order.
  Protocol 1: A) Using a Dynamic Vessel Analyzer, the diameter of a larger retinal vascular arcade arteriole will be recorded for 90 seconds at baseline followed by a similar recording during stimulation with flickering light and a recording during rest, altogether lasting 4.5 minutes. B) Intravenous injection of 0,4 mg regadenoson and repetition of the procedures in step A.
  Protocol 2: The procedures are similar to those of protocol 1 but are performed during breathing of a hypoxic gas mixture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy person (Experimental): The purpose is to investigate the effect of A2A adrenoceptor stimulation using the drug regadenoson (Rapiscan) on the diameter of retinal arterioles during hypoxia in vivo.
  Interventions: Biological: Hypoxia; Drug: Regadenoson

INTERVENTIONS:
Biological: Hypoxia — The purpose is to test the effect of A2A adrenoceptor stimulation on the diameter of retinal arterioles during hypoxia in vivo
Drug: Regadenoson — The purpose is to test the effect of A2A adrenoceptor stimulation on the diameter of retinal arterioles during hypoxia in vivo
  Other Names: Rapiscan

SUMMARY:
The purpose is to investigate how the adenosine affects the diameter regulation of retinal arterioles during changes in oxygen tension. A deeper understanding of the mechanisms involved in diameter regulation of retinal arterioles during changes in oxygen tension can be used to obtain a more detailed understanding of diseases where changes in the diameter regulation of retinal vessels are involved in the disease pathogenesis and possibly point to new therapeutic options for patients with retinal vascular disease, such as diabetic retinopathy and retinal vein thrombosis.

Preliminary, a routine ophthalmological evaluation, measurement of blood pressure, and electrocardiogram will be preformed to insure that only healthy test persons are included in the study.

The test persons will be randomly allocated to two groups, one group in which protocol 1 is followed by protocol 2, and the other group with the two protocols performed in the reverse order.

Protocol 1: Using the DVA, a video recording will capture the diameter of retinal vessels and the changes occurring during stimulation with flickering light. The recording lasts 4.5 minutes and is preformed before and after intravenous injection of adenosine.

Protocol 2: The procedures are similar to those of protocol 1 but are performed during breathing of a gas mixture with a reduced oxygen tension to 12,5 %, which results in a reduced oxygen saturation in the blood to 85-90 %.

DETAILED DESCRIPTION:
Background:

Occlusion of the retinal vessels leading to retinal ischaemia and hypoxia is an important element in the pathophysiology of the major vision threatening diseases in the Western World. The hypoxic areas release vasodilating factors that induce vasodilatation in adjacent retinal areas in order to increase blood flow and retinal oxygenation. An understanding of the mechanisms underlying this vasodilatation may help identifying new therapeutic principles for modulating retinal blood flow during changes in retinal blood flow secondary to hypoxia and other diseases.

The present study:

Two working hypotheses will be tested: 1) That systemic administration of an A2A adrenoceptor agonist affects retinal blood flow independently of its systemic effects. 2) That the vasodilating effect of A2A adrenoceptor stimulation and the vasodilating effects of systemic hypoxia and increased retinal metabolism induced by flicker stimulation are additive.

Methods:

The diameter of retinal vessels are measured using the Dynamic Vessel Analyser (DVA). This apparatus performs video recordings of the ocular fundus, and the single images in the video sequences are grabbed for computerised analysis. Special software enables calculation of the diameter of the vessel on the basis of the distance between the vessel borders. The fact that images are grabbed real time (25 times per second) allows the detection of immediate diameter changes when the retinal metabolism is increased by exposure to flickering light (metabolic autoregulation).

The A2A adrenoceptor agonist regadenoson is administered during continuous ECG monitoring as a single intravenous injection of 400 micrograms (5 ml) in an antecubital vein. No dose adjustments are necessary for body weight, age, renal og hepatic impairment. Due to a potential ischaemic effect of regadenoson, only persons with no history of arterial hypertension or cardiac disease and with normal blood pressure and ECG will be included.

The experiments will be performed during breathing of ambient air and after 10 minutes of breathing air containing 12.5% oxygen (corresponding to the saturation at an altitude of 4100 m), which induces a decline in the arterial oxygen saturation resulting in dilatation of retinal vessels.

Experimental design:

The project will be conducted as an open controlled interventional study performed on two days separated by at least one day. Initial a routine ophthalmological evaluation with a slit lamp examination, measurement of the intraocular pressure and ophthalmoscopy, supplemented with a measurement of central retinal thickness using optical coherence tomography scanning will be preformed as will measuring of ECG and blood pressure to make sure only healthy test persons are included.

The test persons will be randomly allocated to two groups, one group in which protocol 1 is followed by protocol 2, and the other group with the two protocols performed in the reverse order.

Protocol 1:

A) Using the DVA, the diameter of a larger retinal vascular arcade arteriole will be recorded for 90 seconds at baseline followed by a similar recording during stimulation with flickering light and a recording during rest, altogether lasting 4.5 minutes B) Intravenous injection of 0,4 mg regadenoson and repetition of the procedures in step A

Protocol 2:

The procedures are similar to those of protocol 1 but are performed during breathing of a hypoxic gas mixture.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-35
* Healthy, both current and prior
* Normal echocardiogram
* Signed and informed consent

Exclusion Criteria:

* Former or current cardiovascular disease or high blood pressure
* Lung diseases incl. asthma or chronic obstructive pulmonary disease (COPD)
* Known eye disease or previously treated for an eye disease, particularly glaucoma and cataracts
* People taking medication, except birth control pills
* Persons who have or who have had epilepsy
* Pregnant or breast-feeding women
* Allergies to the constituent substance of the medication used in the study

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Diameter responses of retinal arterioles | 11 minutes
  The main outcome variable of the DVA is the width measurement of the selected vessel(s), expressed in units of measurement (UM). In a normal Gullstrand eye, 1 UM is equivalent to 1 µm. For the stimulation with flicker light, the outcome is defined as the percent change from baseline.

SECONDARY OUTCOMES:
Blood pressure | The blood pressure is measured during the last 40 seconds in each phase using an oscillometric technique on the left arm.
  mmHg
Systemic arterial saturation | The systemic arterial saturation is registered at the beginning and half way through each examination phase and during the 2 min break where the drug Regadenoson is injected.
  Percentage
Intraocular pressure | The intraocular pressure is measured before and after the drug administration (time point 280 and 350 sec) and after the second DVA examination is terminated (time point 670 sec).
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Toke Bek, Chair, Study Chair — Main supervisor
Locations (1):
- Department of Ophthalmology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The project results will be published in recognized international journals. Both positive, negative and inconclusive results will be published.